CLINICAL TRIAL: NCT03113630
Title: Efficacy of Different Interaction Devices Using Virtual Task in Amyotrophic Lateral Sclerosis
Brief Title: Virtual Task in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105/15
Record Dates: First submitted 2017-04-02; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Virtual Reality Exposure Therapy; User-Computer Interface; Rehabilitation; Motor Activity
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Acquisition on TouchScreen (Experimental): Subjects practice the task and retention TouchScreen, transfer 1 on LeapMotion and transfer 2 on Kinect
  Interventions: Device: Acquisition on TouchScreen
- Acquisition on Kinect (Experimental): Subjects practice the task and retention Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Interventions: Device: Acquisition on Kinect
- Acquisition on LeapMotion (Experimental): Subjects practice the task and retention LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Interventions: Device: Acquisition on LeapMotion
- Acquisition on TouchScreen Control Group (Active Comparator): Subjects practice the task and retention TouchScreen, transfer 1 on LeapMotion and transfer 2 on Kinect
  Interventions: Device: Acquisition on TouchScreen Control Group
- Acquisition on Kinect Control Group (Active Comparator): Subjects practice the task and retention Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Interventions: Device: Acquisition on Kinect Control Group
- Acquisition on LeapMotion Control Group (Active Comparator): Subjects practice the task and retention LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Interventions: Device: Acquisition on LeapMotion Control Group

INTERVENTIONS:
Device: Acquisition on TouchScreen — Participants performed acquisition and retention on TouchScreen, transfer 1 on Kinect and transfer 2 on LeapMotion.
  Arms: Acquisition on TouchScreen
Device: Acquisition on Kinect — Participants performed acquisition and retention on Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Arms: Acquisition on Kinect
Device: Acquisition on LeapMotion — Participants performed acquisition and retention on LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Arms: Acquisition on LeapMotion
Device: Acquisition on TouchScreen Control Group — Participants performed acquisition and retention on TouchScreen, transfer 1 on Kinect and transfer 2 on LeapMotion.
  Arms: Acquisition on TouchScreen Control Group
Device: Acquisition on Kinect Control Group — Participants performed acquisition and retention on Kinect, transfer 1 on TouchScreen and transfer 2 on LeapMotion.
  Arms: Acquisition on Kinect Control Group
Device: Acquisition on LeapMotion Control Group — Participants performed acquisition and retention on LeapMotion, transfer 1 on TouchScreen and transfer 2 on Kinect.
  Arms: Acquisition on LeapMotion Control Group

SUMMARY:
Thirty individuals with ALS (18 men and 12 women, mean age 59 years, range 44-74 years), and 30 healthy controls matched for age and gender, participated. Individuals with ALS and from the control group were randomly divided into three groups, each using a different communication device systems (Kinect®, Leap Motion Controller® or touchscreen) to perform two task phases (acquisition and retention). Performance was then explored in a third phase (transfer) by switching devices (two transfers); so that, all groups had contact with all communication interfaces.

DETAILED DESCRIPTION:
Participants A total of 60 individuals participated in this study, 30 individuals with ALS (18 men and 12 women, mean age 59 years, range 44-74 years) and 30 healthy individuals who formed the control group, which were (equally) matched individually for age and gender with ALS group.

Rating scales For clinical characteristics of the participants, the scales of functional assessment, fatigue and quality of life were applied. As a functional assessment tool, the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS - R) was used, validated in Brazilian individuals with ALS which allows monitoring of symptoms and limitations of daily living activities. To evaluate fatigue during the execution of tasks, were used the Fatigue Severity Scale (FSS) and for the assessment of quality of life, were used the Amyotrophic Lateral Sclerosis Assessment Questionnaire in the Portuguese Language (ALSAQ-40/BR), which is also validated for the Brazilian population with ALS.

Protocol Subjects were randomly divided into three groups, using different interfaces for the acquisition of movement. The description of the task and the RV interfaces that were used are described as follows.

Task Participants performed a task to test communication devices developed by the Information Systems Team at the University of São Paulo. The task was set up as a game in which the goal was to reach as many bubbles displayed on an 11-inch computer monitor, forming seven rows and 18 columns with a total of 126 bubbles. This required individuals to be able to use a range as is typically required in communication systems. The task was divided into two phases: (1) the first phase was characterized by identification of dexterity zone or range of reach, in which the subject had to touch ("burst") the largest possible number of bubbles (changing bubble color from blue to gray) in a set time of 30 seconds, identifying the range zone; (2) the second phase was characterized as the persecution stage, at this time the researcher defined a central bubble (usually chosen in the center of the skill area, on the bottom line), which changed the color to red. From this moment the individual pursued random bubbles that appeared in their range zone, alternating with a return to the central bubble. This phase was carried out for 30 seconds. To motivate, the task randomly provided bubbles outside the range zone and generated a greater challenge to the individual. The software generated information of the coordinates x, y (row and column) where the bubble was touched and the time the bubble was touched. During task execution, the participant received feedback of the number of bubbles touched, the remaining playing time and the total number of points obtained in attempts, thus observing the performance of the participants.

Interfaces To perform the task were used 3 different interfaces: two interfaces without physical contact, being the Kinect® for Windows from Microsoft, composed of a traditional RGB camera and an infrared depth sensor (IR) and LMC®, characterized as a small motion sensor that demonstrated robustness to measure the movements of the hand and fingers. The interface with physical contact, the touchscreen, was the computer screen itself, where individuals touched the screen in order to burst the bubbles, performing the task. It is noteworthy that the touchscreen is a sensitive interface, employed through pressure, created in order to interact with digital information, found in a majority of modern consumer electronics, mainly computers, tablets and mobile phones.

Procedures and design Individuals who participated in the study gave written informed consent and then were sent to a reserved and quiet room to perform the tasks only in the presence of the researcher. The computer monitor was positioned on a table in front of the participants. The chair was adjusted in accordance with the size and need of the individual, with a footrest available if needed. For wheelchair users, their own wheelchair was used. After the necessary adjustments to perform the task, questionnaires and functional assessment scales were applied; then the researcher provided verbal instructions and performed a demonstration of interfaces according to each task (Kinect® for Windows, LMC® or touchscreen). Subjects were instructed to use the dominant hand (i.e., the least affected side) for all interfaces used during the game.

For the acquisition phase a target was set of 300 bubbles to be touched in the definition phase of the dexterity zone. There were 126 bubbles presented during each attempt; therefore it took at least three attempts to reach the proposed goal. Soon after the step establishing the dexterity zone, the researcher defined the central bubble and began the stage of chase area. In addition to the acquisition phase, all groups performed a retention test after 5 minutes with the completion of only one attempt. After the retention test, two transfer tests with the change of interfaces were performed.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with ALS defined according to the revised classification of El Escorial;
* individuals who regularly attended the Neuromuscular Disease Research Sector (SIDNM) of the Federal University of São Paulo

Exclusion Criteria:

* individuals who had other diagnosis of neuromuscular disease such as: progressive muscular atrophy (PMA), progressive bulbar paralysis (PBP), primary lateral sclerosis (PLS);
* individuals associated with other neurodegenerative diseases;
* those presenting established functional disability that would prevent the completion of the task.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Motor performance improvement in a virtual Timing Coincident task, comparing performance between LeapMotion, TouchScreen and Kinect. | 3 months
  Analysis of the motor performance using a virtual Coincident timing task in different devices to compare wether a task with or without contact promote better performance for people with Amyotrophic Lateral Sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trevizan IL, Silva TD, Dawes H, Massetti T, Crocetta TB, Favero FM, Oliveira ASB, de Araujo LV, Santos ACC, de Abreu LC, Coe S, Monteiro CBM. Efficacy of different interaction devices using non-immersive virtual tasks in individuals with Amyotrophic Lateral Sclerosis: a cross-sectional randomized trial. BMC Neurol. 2018 Dec 17;18(1):209. doi: 10.1186/s12883-018-1212-3. PMID 30558556